CLINICAL TRIAL: NCT02330562
Title: Phase 1, Multicenter, Open-label, Dose-escalation, Combination Study of Marizomib and Bevacizumab in Bevacizumab-Naïve Subjects With WHO Grade IV Malignant Glioma Followed by Phase 2 Studies of Single Agent Marizomib and Combination Marizomib and Bevacizumab, and Phase 1 Dose-Escalation Study of Enterally-administered Marizomib With Bevacizumab
Brief Title: Stage 1: Marizomib + Bevacizumab in WHO Gr IV GBM; Stage 2: Marizomib Alone; Stage 3: Combination of Marizomib and Bevacizumab
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Collaborators: Triphase Research and Development III Corp. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRZ-108
Record Dates: First submitted 2014-12-20; First posted 2015-01-05 (Estimated); Results first posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-05

CONDITIONS: Malignant Glioma; Glioblastoma
Keywords: Marizomib; Bevacizumab; Avastin; Grade IV malignant glioma; proteasome inhibitor; glioblastoma; brain tumor; malignant glioma; brain cancer; gliosarcoma; BEV
MeSH Terms: conditions — Glioma; Glioblastoma; Brain Neoplasms; Gliosarcoma | interventions — marizomib; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Phase 1: MRZ + BEV; Phase 2: MRZ alone (Experimental): Part1-Phase1: MRZ 10 minute IV infusion on Days 1, 8, and 15 plus BEV IV infusion on Days 1 and 15 of each 28-day cycle.
  Part2-Phase2: MRZ 10 minute IV infusion administered on Days 1, 8, and 15 of each 28-day cycle.
  Part3-Phase2: All subjects will receive IV MRZ infusion and IV BEV infusion. MRZ will be administered as a 10-minute, IV infusion on Days 1, 8, and 15 of every 28-day cycle using intra-patient dose escalation. Starting dose will be 0.8 mg/m2.
  Part4- Phase1: All subjects will receive MRZ enterally by NG tube as a bolus on Days 1, 8 and 15 of the first 28-day cycle and BEV IV infusion on Day 15 of the first 28-day cycle. For subsequent 28-day treatment cycles, MRZ will be administered as an IV at the recommended dose and schedule determined in Part 1, with BEV IV on Days 1 and 15.
  Part5-Phase1: All subjects will receive IV MRZ infusion and IV BEV infusion. MRZ will be administered as a 10-minute, IV infusion at 0.8 mg/m2 on Days 1, 8, and 15 of every 28-day cycle 0.8 mg/m2
  Interventions: Drug: MRZ; Drug: BEV

INTERVENTIONS:
Drug: MRZ — MRZ dosing in Phase 1 to range from 0.55 to 0.8 mg/m2. Dose Escalation: MRZ dose-escalation will occur using a standard 3+3 study design.
  The RP2D of MRZ (0.8.mg/m2) will be used in a two stage design, with fifteen response-evaluable patients entered in the first stage. If 1 or more responses are observed at the MRZ RP2D, then the second stage will be implemented with an additional 15 response-evaluable patients treated.
  Other Names: Marizomib, CC-92763, NPI-0052
Drug: BEV — BEV 10 mg/kg IV infusion administered for all cohorts in Phase 1 only.
  Other Names: Avastin, Bevacizumab

SUMMARY:
This is a Phase 1/2 clinical trial to evaluate a new combination of drugs, marizomib (MRZ) and bevacizumab (BEV; Avastin®), for the treatment of WHO Grade IV malignant glioma. The study population includes subjects who are in first or second relapse and who have not previously received any bevacizumab or other anti-angiogenic agent or proteasome inhibitor for treatment of malignant glioma. Part 1 Phase 1 evaluates the combination of MRZ and BEV, while Part 2 Phase 2 evaluates single-agent MRZ. Part 3 (Phase 2) includes a combination MRZ using intra-patient dose escalation, and BEV at a fixed dose. Part 4 Phase 1 evaluates MRZ through enteral administration, and BEV at a fixed dose. Part 5 Phase 1 evaluates the repeat-dose pharmacokinetics of MRZ administered IV with ECG.

DETAILED DESCRIPTION:
One of the few treatment options currently FDA approved for recurrent WHO Grade IV malignant glioma is BEV. Additional treatment options are needed for these subjects. Published literature indicates that targeting the proteasome in glioma cells has shown significant anti-tumor activity.

MRZ is a novel, second generation proteasome inhibitor that prevents the breakdown of proteins involved in signal transduction which blocks growth and survival of cancer cells. In-vitro studies of multiple glioma cell lines were highly sensitive to MRZ. MRZ had relatively little effect on neural stem/progenitor cells suggesting minimal neurotoxicity while significantly affecting both malignant glioma stem cells and glioma cell lines.

Parts 1 and 2 of this trial have been completed with the Recommended Part 3 (Phase 2) Dose established at 0.8 mg/m2. Part 3 of this trial is enrolling at the MRZ RP2D determined in Phase 1 to assess the combination of MRZ and BEV activity and safety.

Parts 1, 2, 3 and 4 of this trial have been completed with the Recommended Dose established at 0.8 mg/m2. Part 5 of this trial is enrolling.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign and date an informed consent document prior to any study related assessments/procedures are conducted.
2. Males and females at least 18 years of age at the time of signing of the informed consent document.
3. All subjects must have histologic evidence of G4 MG (including glioblastoma and gliosarcoma) and radiographic evidence of recurrence or disease progression (defined as either a greater than 25% increase in the largest bidimensional product of enhancement, a new enhancing lesion, or significant increase in T2 FLAIR).
4. Subjects must have previously completed standard radiation therapy and been exposed to temozolomide. Patients must be in first or second relapse.
5. No prior treatment with MRZ or any other proteasome inhibitors or any other anti-angiogenic agents.
6. No investigational agent within 4 weeks prior to first dose of study drug.
7. At least 4 weeks from surgical resection and 12 weeks from end of radiotherapy prior to enrollment in this study, unless relapse is confirmed by tumor biopsy or new lesion outside of radiation field, or if there are two MRIs confirming progressive disease that are 8 weeks apart.
8. Subjects with a history of seizures must be on a stable dose of anti-epileptic drugs (AEDs) and without seizures for 14 days prior to enrollment in patients enrolled prior to Amendment 2. Subjects enrolled after Amendment 2 is approved with a history of seizures must be on a stable dose of anti-epileptic drugs (AEDs) for 7 days prior to enrollment.
9. All AEs resulting from prior chemotherapy, surgery, or radiotherapy, must have resolved to at least NCI-CTCAE (v. 4.03) Grade 1 (except for laboratory parameters outlined below).
10. Laboratory results within 7 days prior to MRZ administration (transfusions and/or growth factor support may not be used to meet this criteria):

    * Platelet count at least 100,000/mm3
    * Hemoglobin at least 9 g/dL
    * Absolute neutrophil count (ANC) at least 1,500/mm3
    * Serum bilirubin at least 1.5 × upper limit of normal (ULN) or at least 3 × ULN if Gilbert's disease is documented
    * Aspartate transaminase (AST) at least 2.5 ULN
    * Alanine transaminase (ALT) at least 2.5 ULN
    * Serum creatinine at least 1.5 × ULN
    * Urine protein: creatinine ratio ≤ 1.0 at screening
11. Karnofsky Performance Status (KPS) score at least 70%.
12. For women of child-bearing potential and for men with partners of child-bearing potential, subject must agree to take contraceptive measures for duration of treatments and 6 months after the last dose of BEV. A female subject of childbearing potential (FCBP) is a female who: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (ie, has had menses at any time in the preceding 24 consecutive months).
13. Willing and able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

1. Co-medication that may interfere with study results, eg, immuno-suppressive agents other than corticosteroids. (Steroid therapy for control of cerebral edema is allowed at the discretion of the Investigator. Subjects should be on a stable dose of steroids for at least 1 week prior to first dose of MRZ. Co-medications must not be taken for 2 hours prior to and up to 2 hours after enteral administration of MRZ (Part 4 Phase 1).
2. Evidence of CNS hemorrhage on baseline MRI or CT scan (except for post-surgical, asymptomatic Grade 1 hemorrhage that has been stable for at least 3 months for subjects enrolled prior to Amendment 2 and for at least 4 weeks in subjects enrolled after Amendment 2 is approved).
3. History of thrombotic or hemorrhagic stroke or myocardial infarction within 6 months.
4. Chemotherapy administered within 4 weeks (except 6 weeks for nitrosoureas, 12 weeks for an implanted nitrosoureas wafer, and 1 week from metronomic chemotherapy, such as daily temozolomide and etoposide) prior to Day 1 of study treatment, unless the subject has recovered from all expected toxicities from the chemotherapy.
5. (Part 4 Phase 1) Recent nasal or esophageal surgery, history of GI-related medical conditions, or any other condition which, in the opinion of the investigator, would interfere or cause undue risk with insertion of NG tube or enteral administration of marizomib through the NG tube.
6. Pregnancy or breast feeding.
7. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring IV antibiotics & psychiatric illness/social situations that would limit compliance with study requirements, or disorders associated with significant immunocompromised state.
8. Known previous/current malignancy requiring treatment within ≤ 3 years except for cervical carcinoma in situ, squamous or basal cell skin carcinoma, and superficial bladder carcinoma.
9. Any comorbid condition that confounds the ability to interpret data from the study as judged by the Investigator or Medical Monitor.

   BEV-Specific Concerns (Note: These exclusion criteria apply to the Part 2 Phase 2 portion of the study even though BEV is not administered so that the subject populations among Part 1, Part 2, Part 3, Part 4, and Part 5 are similar):
10. Any prior history of hypertensive crisis or hypertensive encephalopathy.
11. Systolic blood pressure (BP) > 150 mmHg or diastolic BP > 100 mmHg.
12. Unstable angina.
13. New York Heart Association Grade ≥ II congestive heart failure.
14. History of myocardial infarction within 6 months.
15. Subjects with mean QTcF interval > 500 ms.
16. Clinically significant peripheral vascular disease.
17. Evidence of bleeding diathesis, coagulopathy as documented by an elevated (≥ 1.5 x ULN) prothrombin time (PT), partial thromboplastin time (PTT), or bleeding time. The use of full-dose oral or parenteral anticoagulants is permitted as long as the PT or aPTT is within therapeutic limits (according to the medical standard of the enrolling institution) and the subject has been on a stable dose of anticoagulants for at least 2 weeks prior to the first study treatment.
18. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1 or anticipation of need for major surgical procedure during course of the study.
19. Minor surgical procedures, fine needle aspirations or core biopsies within 7 days prior to Day 1.
20. History of abdominal fistula, GI perforation, or intra-abdominal abscess within 6 months prior to Day 1.
21. Serious, non-healing wound, ulcer, or bone fracture requiring surgical intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2015-04-15 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ileana Elias, MD, Study Director — Celgene Corporation
Locations (5):
- United States (4):
  - University of Californai, Irvine, Orange, California
  - John Wayne Cancer Institute, Santa Monica, California
  - Weill Cornell Medical College, New York, New York
  - Duke Univ Medical Center, Durham, North Carolina
- Princess Margaret Hospital, Medical Oncology, Toronto, Ontario, Canada

REFERENCES:
- See also: UC Irvine Health Comprehensive Brain Tumor Program — http://www.ucirvinehealth.org/medical-services/brain-tumor-program/
- See also: The Preston Robert Tisch Brain Tumor Center at Duke University Medical Center — http://www.cancer.duke.edu/btc/
- See also: Brain Tumor Center at New York-Presbyterian Hospital/Weill Cornell Medical Center — http://weillcornellbrainandspine.org/brain-tumor-center
- See also: John Wayne Cancer Institute at Providence Saint John's Health Center — http://california.providence.org/john-wayne/

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1 Cohort 1: Marizomib 0.55 mg/m2 on Days 1,8, and 15 of each 28-day cycle + Bevacizumab 10 mg/Kg on Days 1 and 15 of each 28-day cycle
- Part 1 Cohort 2: Marizomib 0.7 mg/m2 on Days 1,8, and 15 of each 28-day cycle + Bevacizumab 10 mg/Kg on Days 1 and 15 of each 28-day cycle
- Part 1 MTD + Dose Expansion Cohort: Marizomib 0.8 mg/m2 on Days 1,8, and 15 of each 28-day cycle + Bevacizumab 10 mg/Kg on Days 1 and 15 of each 28-day cycle.
  MTD = Maximum Tolerated Dose
- Part 2 Cohort: Marizomib 0.8 mg/m2 on Days 1, 8, and 15 of each 28-day cycle
- Part 3 Cohort 1: Marizomib 0.8 mg/m2 on Days 1,8, and 15 of each 28-day cycle + Bevacizumab 10 mg/Kg on Days 1 and 15 of each 28-day cycle. Based on presence of dose-limiting adverse events, participants did not escalate Marizomib to a dose of 1.0 mg/m2
- Part 3 Cohort 2: Marizomib 0.8 mg/m2 on Days 1,8, and 15 of each 28-day cycle + Bevacizumab 10 mg/Kg on Days 1 and 15 of each 28-day cycle. Based on lack of dose-limiting adverse events for at least 1 cycle, participants were allowed to escalate Marizomib to a dose of 1.0 mg/m2
- Part 4 Cohort 1: Marizomib 0.075 mg/m2 enterally-administered on Days 1,8, and 15 of each 28-day cycle + Bevacizumab 10 mg/Kg on Days 1 and 15 of each 28-day cycle. From Cycle 2, Marizomib was administered at a dose of 0.8 mg/m2 IV
- Part 4 Cohort 2: Marizomib 0.225 mg/m2 enterally-administered on Days 1,8, and 15 of each 28-day cycle + Bevacizumab 10 mg/Kg on Days 1 and 15 of each 28-day cycle. From Cycle 2, Marizomib was administered at a dose of 0.8 mg/m2 IV
- Part 4 Cohort 3: Marizomib 0.675 mg/m2 enterally-administered on Days 1,8, and 15 of each 28-day cycle + Bevacizumab 10 mg/Kg on Days 1 and 15 of each 28-day cycle. From Cycle 2, Marizomib was administered at a dose of 0.8 mg/m2 IV
- Part 4 Cohort 4: Marizomib 1.0 mg/m2 enterally-administered on Days 1,8, and 15 of each 28-day cycle + Bevacizumab 10 mg/Kg on Days 1 and 15 of each 28-day cycle. From Cycle 2, Marizomib was administered at a dose of 0.8 mg/m2 IV
- Part 4 Cohort 5: Marizomib 1.35 mg/m2 enterally-administered on Days 1,8, and 15 of each 28-day cycle + Bevacizumab 10 mg/Kg on Days 1 and 15 of each 28-day cycle. From Cycle 2, Marizomib was administered at a dose of 0.8 mg/m2 IV
Period: Overall Study
Arm/Group | Part 1 Cohort 1 | Part 1 Cohort 2 | Part 1 MTD + Dose Expansion Cohort | Part 2 Cohort | Part 3 Cohort 1 | Part 3 Cohort 2 | Part 4 Cohort 1 | Part 4 Cohort 2 | Part 4 Cohort 3 | Part 4 Cohort 4 | Part 4 Cohort 5
Started | 6 | 3 | 27 | 30 | 31 | 10 | 1 | 1 | 1 | 5 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 3 | 27 | 30 | 31 | 10 | 1 | 1 | 1 | 5 | 6
Not completed — Adverse Event | 0 | 0 | 3 | 0 | 3 | 1 | 0 | 0 | 0 | 1 | 1
Not completed — Participant decision | 1 | 0 | 4 | 1 | 5 | 2 | 0 | 0 | 0 | 3 | 0
Not completed — Disease progression | 5 | 3 | 20 | 28 | 23 | 7 | 1 | 1 | 1 | 0 | 5
Not completed — Other reasons | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 Cohort 1 | Part 1 Cohort 2 | Part 1 MTD + Dose Expansion Cohort | Part 2 Cohort | Part 3 Cohort 1 | Part 3 Cohort 2 | Part 4 Cohort 1 | Part 4 Cohort 2 | Part 4 Cohort 3 | Part 4 Cohort 4 | Part 4 Cohort 5 | Total
Number analyzed (Participants) | 6 | 3 | 27 | 30 | 31 | 10 | 1 | 1 | 1 | 5 | 6 | 121
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 3 | 20 | 23 | 25 | 7 | 0 | 1 | 1 | 5 | 6 | 97
  >=65 years | 0 | 0 | 7 | 7 | 6 | 3 | 1 | 0 | 0 | 0 | 0 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 12 | 13 | 14 | 7 | 1 | 1 | 0 | 4 | 2 | 55
  Male | 5 | 3 | 15 | 17 | 17 | 3 | 0 | 0 | 1 | 1 | 4 | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 5 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 8
  Not Hispanic or Latino | 6 | 3 | 22 | 28 | 31 | 9 | 1 | 1 | 1 | 5 | 6 | 113
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 2 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 4
  White | 5 | 3 | 21 | 27 | 27 | 9 | 1 | 1 | 1 | 5 | 6 | 106
  More than one race | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Objective Response Rate (ORR) - Part 2 Cohort
Description: Radiographic ORR is defined as the percentage of participants achieving a Complete Response (CR) or Partial Response (PR), as assessed by the investigator, according to RANO 2010 criteria.
  Tumor response assessment was conducted every 2 cycles of study therapy. 95% confidence interval from exact binomial distribution (Clopper-Pearson method).
Time Frame: From first dose to end of study treatment (up to approx. 48 weeks)
Population: All treated participants in Part 2 Cohort
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Part 2 Cohort
Number analyzed (Participants) | 30
Percent of participants | 3.3 [0.1 to 17.2]

2. Primary Outcome: Overall Survival (OS) - Part 3 Cohorts
Description: OS is defined as time from the date of the first dose of study drug to date of death due to any cause. Participants who are alive will be censored at the last follow up visit
Time Frame: From first dose to death, assessed up approx. 42 weeks
Population: All treated participants in Part 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 3 Cohort 1 | Part 3 Cohort 2
Number analyzed (Participants) | 31 | 10
Months | 8.3 [4.8 to 11.3] | 7.5 [3.5 to 12.9]

3. Secondary Outcome: Number of Participants Experiencing Adverse Events
Description: Number of subjects experiencing at least 1 Treatment-Emergent Adverse Event (TEAE) within the timeframe specified.
  For Part 4, data are presented separately for Cycle 1 (when Marizomib was enterally-administered) and for Cycles 2 and subsequent cycles (when Marizomib was administered IV)
Time Frame: From first dose to 28 days following last dose (up to approx. 72 weeks for Part 1, approx. 52 weeks for Part 2, approx. 46 weeks for Part 3, and approx. 37 weeks for Part 4)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Groups:
- Part 4 Cohort 1 - Cycle 1: Marizomib 0.075 mg/m2 enterally-administered on Days 1,8, and 15 + Bevacizumab 10 mg/Kg on Days 1 and 15
- Part 4 Cohort 2 - Cycle 1: Marizomib 0.225 mg/m2 enterally-administered on Days 1,8, and 15 + Bevacizumab 10 mg/Kg on Days 1 and 15
- Part 4 Cohort 3 - Cycle 1: Marizomib 0.675 mg/m2 enterally-administered on Days 1,8, and 15 + Bevacizumab 10 mg/Kg on Days 1 and 15
- Part 4 Cohort 4 - Cycle 1: Marizomib 1.0 mg/m2 enterally-administered on Days 1,8, and 15 + Bevacizumab 10 mg/Kg on Days 1 and 15
- Part 4 Cohort 5 - Cycle 1: Marizomib 1.35 mg/m2 enterally-administered on Days 1,8, and 15 + Bevacizumab 10 mg/Kg on Days 1 and 15
- Part 4 All Cohorts - Cycles 2 and Subsequent: Marizomib at different dosage IV-administered on Days 1,8, and 15 of each 28-day cycle + Bevacizumab 10 mg/Kg on Days 1 and 15 of each 28-day cycle
Arm/Group | Part 1 Cohort 1 | Part 1 Cohort 2 | Part 1 MTD + Dose Expansion Cohort | Part 2 Cohort | Part 3 Cohort 1 | Part 3 Cohort 2 | Part 4 Cohort 1 - Cycle 1 | Part 4 Cohort 2 - Cycle 1 | Part 4 Cohort 3 - Cycle 1 | Part 4 Cohort 4 - Cycle 1 | Part 4 Cohort 5 - Cycle 1 | Part 4 All Cohorts - Cycles 2 and Subsequent
Number analyzed (Participants) | 6 | 3 | 27 | 30 | 31 | 10 | 1 | 1 | 1 | 5 | 6 | 11
Participants | 6 | 3 | 27 | 30 | 31 | 10 | 1 | 1 | 1 | 5 | 6 | 11

4. Secondary Outcome: Number of Participants Experiencing Serious Adverse Events (SAEs)
Description: Number of subjects experiencing at least 1 Serious Adverse Event (SAE) within the timeframe specified.
  For Part 4, data are presented separately for Cycle 1 (when Marizomib was enterally-administered) and for Cycles 2 and subsequent cycles (when Marizomib was administered IV)
Time Frame: as for outcome 3
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Cohort 1 | Part 1 Cohort 2 | Part 1 MTD + Dose Expansion Cohort | Part 2 Cohort | Part 3 Cohort 1 | Part 3 Cohort 2 | Part 4 Cohort 1 - Cycle 1 | Part 4 Cohort 2 - Cycle 1 | Part 4 Cohort 3 - Cycle 1 | Part 4 Cohort 4 - Cycle 1 | Part 4 Cohort 5 - Cycle 1 | Part 4 All Cohorts - Cycles 2 and Subsequent
Number analyzed (Participants) | 6 | 3 | 27 | 30 | 31 | 10 | 1 | 1 | 1 | 5 | 6 | 11
Participants | 1 | 0 | 12 | 10 | 14 | 5 | 0 | 0 | 0 | 0 | 2 | 4

5. Secondary Outcome: Number of Participants Experiencing Dose-Limiting Toxicity (DLT)
Description: Number of subjects experiencing at least 1 DLT event within the timeframe specified.
  DLT is defined as the occurrence of any of the following AEs related to one of the drugs or the combination observed during Cycle 1, using NCI-CTCAE (v 4.03):
  * ≥ Grade 3 thrombocytopenia or Grade 2 thrombocytopenia with bleeding.
  * Grade 4 neutropenia or anemia lasting for more than 4 days.
  * Febrile neutropenia.
  * Any ≥ Grade 2 neurological event lasting more than 4 days.
  * Grade 3 or 4 non-hematologic toxicity (excluding alopecia), lasting for more than 4 days despite adequate supportive therapy or preventing the next scheduled dose from being administered within 4 days of scheduled day; for ≥ Grade 3 fatigue to be considered a DLT, it must be present for more than 7 days.
  For Part 4, data are presented separately for Cycle 1 (when Marizomib was enterally-administered) and for Cycles 2 and subsequent cycles (when Marizomib was administered IV).
  DLT was assessed only for Part 1 and Part 4 cohorts.
Time Frame: From first dose to 28 days first dose (during Cycle 1 of study treatment)
Population: All treated participants in Part 1 and Part 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Cohort 1 | Part 1 Cohort 2 | Part 1 MTD + Dose Expansion Cohort | Part 4 Cohort 1 - Cycle 1 | Part 4 Cohort 2 - Cycle 1 | Part 4 Cohort 3 - Cycle 1 | Part 4 Cohort 4 - Cycle 1 | Part 4 Cohort 5 - Cycle 1
Number analyzed (Participants) | 6 | 3 | 27 | 1 | 1 | 1 | 5 | 6
Participants | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1

6. Secondary Outcome: Number of Participants Experiencing Dose-Limiting Adverse Events (DLAEs)
Description: Number of subjects experiencing at least 1 DLAE within the timeframe specified.
  DLAEs are defined as Marizomib-related AEs observed which are:
  * related to disturbances in the cerebellum (ie, ataxia, dizziness, dysarthria, fall, gait disturbances) plus hallucinations of any grade
  * any other AEs of Grade ≥ 2. DLAEs were assessed only for Part 3 cohorts.
Time Frame: From first dose to 28 days following last dose (up to approx. 46 weeks)
Population: All treated participants in Part 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part 3 Cohort 1 | Part 3 Cohort 2
Number analyzed (Participants) | 31 | 10
Participants | 31 | 10

7. Secondary Outcome: Radiographic Objective Response Rate (ORR)
Description: Radiographic ORR is defined as the percentage of participants achieving a Complete Response (CR) or Partial Response (PR), as assessed by the investigator, according to RANO 2010 criteria.
  Tumor response assessment was conducted every 2 cycles of study therapy. 95% confidence interval from exact binomial distribution (Clopper-Pearson method).
  Radiographic ORR was assessed for Part 1 and Part 3 cohorts
Time Frame: From first dose to end of study treatment (up to approx. 68 weeks for Part 1, and approx. 42 weeks for Part 3)
Population: All treated participants with available measurements
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Part 1 Cohort 1 | Part 1 Cohort 2 | Part 1 MTD + Dose Expansion Cohort | Part 3 Cohort 1 | Part 3 Cohort 2
Number analyzed (Participants) | 6 | 3 | 25 | 29 | 10
Percent of participants | 50.0 [NA to NA] — Insufficient number of events | 33.3 [NA to NA] — Insufficient number of events | 48.0 [27.8 to 68.7] | 24.1 [10.3 to 43.5] | 20.0 [2.5 to 55.6]

8. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time between start of treatment and first evidence of documented disease progression or death (due to any cause), whichever occurs first. Disease progression will be determined using RANO 2010 criteria as assessed by the investigator.
  PFS was determined using Kaplan-Meier product-limit estimates.
Time Frame: From first dose to disease progression or death, assessed up to approx. 68 weeks for Part 1, approx. 48 weeks for Part 2, approx. 42 weeks for Part 3, and approx. 33 weeks for Part 4
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1 Cohort 1 | Part 1 Cohort 2 | Part 1 MTD + Dose Expansion Cohort | Part 2 Cohort | Part 3 Cohort 1 | Part 3 Cohort 2 | Part 4 Cohort 1 | Part 4 Cohort 2 | Part 4 Cohort 3 | Part 4 Cohort 4 | Part 4 Cohort 5
Number analyzed (Participants) | 6 | 3 | 27 | 30 | 31 | 10 | 1 | 1 | 1 | 5 | 6
Months | 7.3 [NA to NA] — Insufficient number of events | 3.7 [NA to NA] — Insufficient number of events | 3.9 [1.9 to 5.5] | 1.8 [1.5 to 1.9] | 3.5 [2.6 to 3.6] | 2.1 [1.5 to 5.3] | 5.1 [NA to NA] — Insufficient number of events | 2.3 [NA to NA] — Insufficient number of events | 7.4 [NA to NA] — Insufficient number of events | NA [1.8 to NA] — Insufficient number of events | 3.8 [1.9 to NA] — Insufficient number of events

9. Secondary Outcome: Overall Survival (OS)
Description: as for outcome 2
Time Frame: From first dose to death, assessed up to approx. 68 weeks for Part 1, approx. 48 weeks for Part 2, and approx. 33 weeks for Part 4
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1 Cohort 1 | Part 1 Cohort 2 | Part 1 MTD + Dose Expansion Cohort | Part 2 Cohort | Part 4 Cohort 1 | Part 4 Cohort 2 | Part 4 Cohort 3 | Part 4 Cohort 4 | Part 4 Cohort 5
Number analyzed (Participants) | 6 | 3 | 27 | 30 | 1 | 1 | 1 | 5 | 6
Months | 10.4 [NA to NA] — Insufficient number of events | 6.3 [NA to NA] — Insufficient number of events | 10.4 [6.0 to 14.1] | 11.4 [5.5 to 13.0] | 8.3 [NA to NA] — Insufficient number of events | NA [NA to NA] — Insufficient number of events | 14.2 [NA to NA] — Insufficient number of events | NA [7.7 to NA] — Insufficient number of events | 8.7 [1.9 to NA] — Insufficient number of events

ADVERSE EVENTS:
Time Frame: All-cause mortality: from randomization to study completion (up to approximately 73 months) SAEs and Other Adverse Events: from first dose to 28 days following last dose (up to approximately 72 weeks)
Description: All treated participants
Arm/Group | Part 1 Cohort 1 | Part 1 Cohort 2 | Part 1 MTD + Dose Expansion Cohort | Part 2 Cohort | Part 3 Cohort 1 | Part 3 Cohort 2 | Part 4 Cohort 1 | Part 4 Cohort 2 | Part 4 Cohort 3 | Part 4 Cohort 4 | Part 4 Cohort 5
All-Cause Mortality (participants affected / at risk) | 5/6 | 2/3 | 21/27 | 24/30 | 25/31 | 9/10 | 1/1 | 0/1 | 1/1 | 1/5 | 4/6
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/3 | 12/27 | 10/30 | 14/31 | 5/10 | 1/1 | 0/1 | 0/1 | 1/5 | 3/6
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3 | 26/27 | 30/30 | 31/31 | 10/10 | 1/1 | 1/1 | 1/1 | 5/5 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 Cohort 1 (N=6) | Part 1 Cohort 2 (N=3) | Part 1 MTD + Dose Expansion Cohort (N=27) | Part 2 Cohort (N=30) | Part 3 Cohort 1 (N=31) | Part 3 Cohort 2 (N=10) | Part 4 Cohort 1 (N=1) | Part 4 Cohort 2 (N=1) | Part 4 Cohort 3 (N=1) | Part 4 Cohort 4 (N=5) | Part 4 Cohort 5 (N=6)
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Optic nerve disorder (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis perforated (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Wound infection staphylococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 2 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 2
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 3 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Delusion (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 Cohort 1 (N=6) | Part 1 Cohort 2 (N=3) | Part 1 MTD + Dose Expansion Cohort (N=27) | Part 2 Cohort (N=30) | Part 3 Cohort 1 (N=31) | Part 3 Cohort 2 (N=10) | Part 4 Cohort 1 (N=1) | Part 4 Cohort 2 (N=1) | Part 4 Cohort 3 (N=1) | Part 4 Cohort 4 (N=5) | Part 4 Cohort 5 (N=6)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 6 | 6 | 4 | 2 | 0 | 0 | 0 | 2 | 2
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cyanosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Ear congestion (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Cushingoid (Endocrine disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 4
Dry eye (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye disorder (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 1 | 2 | 4 | 3 | 10 | 0 | 0 | 0 | 0 | 0 | 3
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 7 | 10 | 6 | 3 | 0 | 1 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 8 | 7 | 10 | 2 | 0 | 0 | 0 | 3 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 2 | 3 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 3 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faecal incontinence (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 3 | 1 | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 2 | 17 | 11 | 13 | 6 | 1 | 1 | 1 | 5 | 5
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 3 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Tooth disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 16 | 10 | 16 | 6 | 1 | 1 | 1 | 5 | 6
Asthenia (General disorders) | 1 | 0 | 2 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site bruise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Extravasation (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 3 | 2 | 20 | 20 | 24 | 9 | 0 | 0 | 1 | 3 | 5
Gait disturbance (General disorders) | 0 | 1 | 4 | 5 | 15 | 5 | 0 | 0 | 0 | 0 | 2
Influenza like illness (General disorders) | 0 | 0 | 1 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 2
Infusion site erythema (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion site pain (General disorders) | 3 | 1 | 4 | 4 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Infusion site phlebitis (General disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion site reaction (General disorders) | 1 | 1 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 4 | 5 | 1 | 0 | 1 | 1 | 0 | 0 | 1
Pain (General disorders) | 0 | 1 | 2 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 3 | 1 | 5 | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 0 | 7 | 4 | 12 | 3 | 1 | 0 | 0 | 0 | 1
Incision site pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 3 | 1 | 2 | 0 | 1 | 1 | 0 | 1 | 3
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 2 | 3 | 2 | 0 | 1 | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 2 | 5 | 3 | 0 | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 2 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 2 | 5 | 7 | 6 | 0 | 0 | 1 | 0 | 2 | 2
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 2 | 2 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2 | 3 | 3 | 1 | 0 | 0 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 3 | 1 | 0 | 0 | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 6 | 8 | 7 | 1 | 0 | 0 | 0 | 2 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2 | 2 | 4 | 6 | 1 | 0 | 1 | 0 | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 6 | 5 | 0 | 0 | 0 | 0 | 2 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0 | 5 | 8 | 10 | 2 | 0 | 1 | 0 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 6 | 7 | 1 | 0 | 0 | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 3
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 5 | 5 | 10 | 3 | 0 | 0 | 0 | 1 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 1 | 4 | 7 | 6 | 3 | 0 | 0 | 0 | 0 | 3
Ataxia (Nervous system disorders) | 0 | 1 | 7 | 7 | 11 | 2 | 0 | 0 | 1 | 0 | 2
Balance disorder (Nervous system disorders) | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Cerebellar syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 4 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1 | 4 | 4 | 4 | 3 | 1 | 0 | 0 | 1 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 8 | 5 | 12 | 4 | 0 | 0 | 1 | 1 | 3
Dysarthria (Nervous system disorders) | 1 | 0 | 5 | 7 | 9 | 4 | 1 | 0 | 1 | 1 | 2
Dysgeusia (Nervous system disorders) | 0 | 1 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Facial nerve disorder (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Facial paresis (Nervous system disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 4 | 3 | 12 | 14 | 13 | 5 | 1 | 1 | 1 | 1 | 5
Hemianopia homonymous (Nervous system disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 2 | 4 | 3 | 3 | 0 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 7 | 3 | 7 | 0 | 0 | 0 | 0 | 0 | 2
Muscle spasticity (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nystagmus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Paraesthesia (Nervous system disorders) | 1 | 0 | 4 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Partial seizures (Nervous system disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pyramidal tract syndrome (Nervous system disorders) | 0 | 0 | 4 | 3 | 2 | 1 | 0 | 0 | 0 | 1 | 2
Quadranopia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sensory loss (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Sinus headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Tremor (Nervous system disorders) | 1 | 0 | 2 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vasogenic cerebral oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Visual field defect (Nervous system disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 2 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 2
Agitation (Psychiatric disorders) | 0 | 0 | 3 | 0 | 5 | 4 | 0 | 0 | 0 | 0 | 2
Anxiety (Psychiatric disorders) | 3 | 0 | 3 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Confusional state (Psychiatric disorders) | 1 | 0 | 7 | 7 | 16 | 7 | 1 | 0 | 0 | 2 | 3
Depression (Psychiatric disorders) | 2 | 0 | 1 | 2 | 3 | 1 | 0 | 0 | 0 | 1 | 2
Hallucination (Psychiatric disorders) | 0 | 0 | 12 | 12 | 19 | 6 | 1 | 1 | 1 | 1 | 4
Insomnia (Psychiatric disorders) | 1 | 0 | 3 | 13 | 9 | 2 | 0 | 0 | 0 | 0 | 2
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Paranoia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1
Personality change (Psychiatric disorders) | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Glycosuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1 | 3 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 3 | 3 | 5 | 2 | 1 | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 2 | 3 | 0 | 0 | 0 | 0 | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 10 | 1 | 9 | 1 | 0 | 1 | 1 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 3 | 2 | 2 | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 8 | 2 | 2 | 1 | 0 | 0 | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 2 | 2 | 0 | 0 | 0 | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 2 | 2 | 1 | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 3 | 2 | 10 | 3 | 7 | 3 | 0 | 1 | 1 | 1 | 2
Hypotension (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral venous disease (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Vascular pain (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-18): https://cdn.clinicaltrials.gov/large-docs/62/NCT02330562/Prot_SAP_000.pdf